CLINICAL TRIAL: NCT04449029
Title: Phase IIb Multi-Center, Randomised, Partial-Blind Parallel Cohort Study to Assess the Efficacy and Safety of Treatment With GSK3228836 in Participants With Chronic Hepatitis B Virus (B-Clear)
Brief Title: A Study of GSK3228836 in Participants With Chronic Hepatitis B (CHB)
Acronym: B-Clear
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 209668
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-04

CONDITIONS: Hepatitis B
Keywords: Chronic Hepatitis B; GSK3228836; Hepatitis B virus surface antigen; Nucleos(t)ide therapy; Sustained virologic response
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic

STUDY DESIGN:
Intervention Model Description: Participants with CHB will be divided into two different cohorts; participants on stable nucleos(t)ide treatment and participants not currently on nucleos(t)ide therapy. For each cohort, participants will be randomized into one of the 4 different parallel arms to receive treatment.
Who Masked: Participant
Masking Description: Participants will be blinded to the study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1: GSK3228836 300 mg + LD (Experimental): Eligible participants on stable nucleos(t)ide treatment will receive 300 milligrams (mg) GSK3228836 once weekly for 24 weeks along with loading dose (LD) of 300 mg GSK3228836 on Day 4 and Day 11.
  Interventions: Drug: GSK3228836; Drug: Nucleos(t)ide therapy
- Cohort 1: GSK3228836 300 mg + LD/ GSK3228836 150 mg + Placebo (Experimental): Eligible participants on stable nucleos(t)ide treatment will receive 300 mg GSK3228836 once weekly for 12 weeks along with LD of 300 mg GSK3228836 on Day 4 and Day 11 followed by step-down in dose of 150 mg GSK3228836 once weekly for 12 weeks along with placebo to match to maintain participant blinding.
  Interventions: Drug: GSK3228836; Drug: Placebo; Drug: Nucleos(t)ide therapy
- Cohort 1: GSK3228836 300 mg + LD/ Placebo (Experimental): Eligible participants on stable nucleos(t)ide treatment will receive 300 mg GSK3228836 once weekly for 12 weeks along with LD of 300 mg GSK3228836 on Day 4 and Day 11 followed by placebo once weekly for 12 weeks.
  Interventions: Drug: GSK3228836; Drug: Placebo; Drug: Nucleos(t)ide therapy
- Cohort 1: Placebo/ GSK3228836 300 mg + Placebo LD (Experimental): Eligible participants on stable nucleos(t)ide treatment will receive placebo once weekly for 12 weeks followed by 300 mg GSK3228836 once weekly for 12 weeks along with placebo LD to match on Day 4 and Day 11.
  Interventions: Drug: GSK3228836; Drug: Placebo; Drug: Nucleos(t)ide therapy
- Cohort 2: GSK3228836 300 mg + LD (Experimental): Eligible participants not currently on nucleos(t)ide therapy will receive 300 mg GSK3228836 once weekly for 24 weeks along with LD of 300 mg GSK3228836 on Day 4 and Day 11.
  Interventions: Drug: GSK3228836
- Cohort 2: GSK3228836 300 mg + LD/ GSK3228836 150 mg + Placebo (Experimental): Eligible participants not currently on nucleos(t)ide therapy will receive 300 mg GSK3228836 once weekly for 12 weeks along with LD of 300 mg GSK3228836 on Day 4 and Day 11 followed by step-down in dose of 150 mg GSK3228836 once weekly for 12 weeks along with placebo to match to maintain participant blinding.
  Interventions: Drug: GSK3228836; Drug: Placebo
- Cohort 2: GSK3228836 300 mg + LD/ Placebo (Experimental): Eligible participants not currently on nucleos(t)ide therapy will receive 300 mg GSK3228836 once weekly for 12 weeks along with LD of 300 mg GSK3228836 on Day 4 and Day 11 followed by placebo once weekly for 12 weeks.
  Interventions: Drug: GSK3228836; Drug: Placebo
- Cohort 2: Placebo/ GSK3228836 300 mg + Placebo LD (Experimental): Eligible participants not currently on nucleos(t)ide therapy will receive placebo once weekly for 12 weeks followed by 300 mg GSK3228836 once weekly for 12 weeks along with placebo LD to match on Day 4 and Day 11.
  Interventions: Drug: GSK3228836; Drug: Placebo

INTERVENTIONS:
Drug: GSK3228836 — GSK3228836 will be available as a clear colorless to slightly yellow solution for injection at a unit dose strength of 150 mg/mL to be administered subcutaneously once weekly.
Drug: Placebo — Placebo will be available as a clear colorless solution for injection to be administered subcutaneously once weekly.
  Arms: Cohort 1: GSK3228836 300 mg + LD/ GSK3228836 150 mg + Placebo; Cohort 1: GSK3228836 300 mg + LD/ Placebo; Cohort 1: Placebo/ GSK3228836 300 mg + Placebo LD; Cohort 2: GSK3228836 300 mg + LD/ GSK3228836 150 mg + Placebo; Cohort 2: GSK3228836 300 mg + LD/ Placebo; Cohort 2: Placebo/ GSK3228836 300 mg + Placebo LD
Drug: Nucleos(t)ide therapy — Participants receiving nucleos(t)ide therapy upon entry in the study will continue to receive nucleotide therapy for the duration of the study.
  Arms: Cohort 1: GSK3228836 300 mg + LD; Cohort 1: GSK3228836 300 mg + LD/ GSK3228836 150 mg + Placebo; Cohort 1: GSK3228836 300 mg + LD/ Placebo; Cohort 1: Placebo/ GSK3228836 300 mg + Placebo LD

SUMMARY:
Chronic hepatitis B virus (HBV) infection is a significant worldwide medical problem. GSK3228836 demonstrated target engagement in CHB participants who were not on treatment and in CHB participants on stable nucleos(t)ide therapy. This study is intended to evaluate if treatment with GSK3228836 can achieve sustained virologic response (SVR), that is hepatitis B virus surface antigen (HBsAg) less than (<) lower limit of quantitation (LLOQ) and HBV deoxyribonucleic acid (DNA) <LLOQ sustained for 24 weeks post-GSK3228836 treatment end. In addition, the study will also evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic properties of GSK3228836 in the 4 dosing regimens. This study will assess the efficacy and safety of treatment with GSK3228836 in two populations of participants with CHB; participants on stable nucleos(t)ide treatment (Cohort 1) and participants who are not currently on nucleos(t)ide therapy (Cohort 2). For each population, participants will be randomized into one of the 4 different parallel arms to receive treatment. The study will consist of a screening, treatment, and post-treatment follow-up phase. Approximately, 440 participants will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of signing the informed consent.
* Participants who have documented chronic HBV infection greater than equal to (>=6) months prior to screening and not currently on nucleos(t)ide analogue therapy population defined as participants who never received HBV treatment (treatment naive) or must have ended nucleos(t)ide therapy at least 6 months prior to the screening visit; OR Currently receiving stable nucleos(t)ide analogue therapy population defined as no changes to their nucleos(t)ide regimen from at least 6 months prior to screening and with no planned changes to the stable regimen over the duration of the study.
* Plasma or serum HBsAg concentration >100 international units per milliliter (IU/mL).
* Plasma or serum HBV DNA concentration: Participants not currently on nucleos(t)ide analogue therapy, plasma or serum HBV DNA >2000 IU/mL; Participants who are receiving stable nucleos(t)ide analogue therapy must be adequately suppressed, defined as plasma or serum HBV DNA <90 IU/mL.
* ALT for treatment naive participants and for participants who are not currently receiving treatment: ALT <3 times ULN will be included initially if agreed by the independent data monitoring committee (IDMC) after review of safety data, the ALT inclusion criteria may be expanded to include participants with ALT <5 times ULN; ALT less than equal to (<=2) times ULN for participants who are receiving stable nucleos(t)ide analogue therapy.
* Male and/or Female: A male participant is eligible to participate if they agree to the following during the intervention period and for at least 90 days after the last dose of study treatment: Refrain from donating sperm AND be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or Must agree to use contraception/barrier as detailed below: Agree to use a male condom (and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak) when having sexual intercourse with a woman of childbearing potential who is not currently pregnant. A female participant is eligible to participate: If she is not pregnant or breastfeeding AND at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP) OR is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1 percent per year), preferably with low user dependency during the intervention period and for at least 90 days after the last dose of study treatment; A WOCBP must have both a confirmed menstrual period prior to the first dose of study intervention (additional evaluation [e.g., amenorrhea in athletes, birth control] should also be considered) and a negative highly sensitive pregnancy test (urine or serum) within 24 hours before the first dose of study treatment.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Clinically significant abnormalities, aside from chronic HBV infection in medical history (e.g., moderate-severe liver disease other than chronic HBV, acute coronary syndrome within 6 months of screening, major surgery within 3 months of screening, significant/unstable cardiac disease, uncontrolled diabetes, bleeding diathesis or coagulopathy) or physical examination.
* Co-infection with Current or past history of Hepatitis C virus (HCV), Human immunodeficiency virus (HIV), Hepatitis D virus (HDV).
* History of or suspected liver cirrhosis and/or evidence of cirrhosis as determined by both Aspartate aminotransferase (AST)-Platelet Index (APRI) >2 and FibroSure/FibroTest result >0.7. If only one parameter (APRI or FibroSure/FibroTest) result is positive, a discussion with the Medical Monitor is required before inclusion in study is permitted. Regardless of APRI of Fibrosure/FibroTest score, if the participant meets one of the following criteria, they will be excluded from the study: Liver biopsy (i.e., Metavir Score F4); Liver stiffness >12 kilopascals (kPa).
* Diagnosed or suspected hepatocellular carcinoma as evidenced by the following: Alpha-fetoprotein concentration >=200 nanogram per milliliter (ng/mL); If the screening alpha fetoprotein concentration is >=50 ng/mL and <200 ng/mL, the absence of liver mass must be documented by imaging within 6 months before randomization.
* History of malignancy within the past 5 years with the exception of specific cancers that are cured by surgical resection (e.g., skin cancer). Participants under evaluation for possible malignancy are not eligible.
* History of vasculitis or presence of symptoms and signs of potential vasculitis (e.g., vasculitic rash, skin ulceration, repeated blood detected in urine without identified cause) or history/presence of other diseases that may be associated with vasculitis condition (e.g., systemic lupus erythematosus, rheumatoid arthritis, relapsing polychondritis, mononeuritis multiplex).
* History of extrahepatic disorders possibly related to HBV immune conditions (e.g., nephrotic syndrome, any type of glomerulonephritis, polyarteritis nodosa, cryoglobulinemia, uncontrolled hypertension).
* Anti-neutrophil cytoplasmic antibodies (ANCA) at screening by itself won't be an exclusion criterion, but if results are borderline positive or positive: myeloperoxidase-ANCA (MPO-ANCA) (Perinuclear antineutrophil cytoplasmic antibodies [pANCA]) and proteinase 3- ANCA (PR3-ANCA) (Cytoplasmic antineutrophil cytoplasmic antibodies [cANCA]) analysis will be conducted; A discussion with the Medical Monitor will be required to review participant's complete medical history to ensure no past history or current manifestations of a vasculitic/inflammatory/auto-immune condition before inclusion in study is permitted.
* Low complement C3 (C3) at screening by itself won't be an exclusion criterion, but if it is present: A discussion with the Medical Monitor is required to review participant's complete medical history to ensure no past history or current manifestations of vasculitic/inflammatory/auto-immune conditions.
* History of alcohol or drug abuse/dependence: Current alcohol use as judged by investigator to potentially interfere with participant compliance; History of or current drug abuse/dependence as judged by the investigator to potentially interfere with participant compliance. Refers to illicit drugs and substances with abuse potential. Medications that are used by the participant as directed, whether over-the-counter or through prescription, are acceptable and would not meet the exclusion criteria.
* Currently taking, or took within 3 months of screening, any immunosuppressing drugs (e.g., prednisone), other than a short course of therapy (<=2 weeks) or topical/inhaled steroid use.
* Participants for whom immunosuppressive treatment is not advised, including therapeutic doses of steroids, will be excluded.
* Currently taking, or took within 12 months of screening, any interferon-containing therapy.
* Participants requiring anti-coagulation therapies (for example warfarin, Factor Xa inhibitors or anti-platelet agents like clopidogrel).
* The participant has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 5 half-lives (if known) or twice the duration (if known) of the biological effect of the study treatment (whichever is longer) or 90 days (if half-life or duration is unknown).
* Prior treatment with any oligonucleotide or small interfering ribonucleic acid (RNA) (Small interfering RNA [siRNA]) within 12 months prior to the first dosing day.
* Fridericia's QT correction formula (QTcF) >=450 milliseconds (msec) (if single electrocardiogram [ECG] at screening shows QTcF>=450 msec, a mean of triplicate measurements should be used to confirm that participant meets exclusion criterion).
* Laboratory results as follows: Serum albumin <3.5 grams per deciliter (g/dL), Glomerular filtration rate (GFR) <60 milliliter per minute per 1.73 square meter (mL/min /1.73 m^2) as calculated by the Chronic Kidney Disease Epidemiologic Collaboration (CKD-EPI) formula (for Japan, Japanese Society of Nephrology Chronic Kidney Disease Initiative [JSN-CKDI equation]), International normalized ratio (INR) >1.25. Platelet count <140 times 10^9 cells/L, Total bilirubin >1.25 times ULN. For participants with benign unconjugated hyperbilirubinemia with total bilirubin >1.25 times ULN, discussion for inclusion to the study is required with the Medical Monitor, Urine albumin to creatinine ratio (ACR) >=0.03 mg/mg (or >=30 mg/g). In the event of an ACR above this threshold, eligibility may be confirmed by a second measurement. In cases where participants have low urine albumin and low urine creatinine levels resulting in a urine ACR calculation >=0.03 mg/mg (or >=30 mg/g), the investigator should confirm that the participant does not have a history of diabetes, hypertension or other risk factors that may affect renal function and discuss with the Medical Monitor, or designee.
* History of/sensitivity to GSK3228836 or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (97):
- United States (7):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Richmond, Virginia
- Argentina (2):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Buenos Aires
- Bulgaria (2):
  - GSK Investigational Site, Sliven
  - GSK Investigational Site, Sofia
- Canada (7):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
  - GSK Investigational Site, Québec
- China (6):
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Chongqing, Sichuan
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Shanghai
- France (6):
  - GSK Investigational Site, Clichy
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Strasbourg
- Germany (4):
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Pokfulam, Hong Kong
- Italy (2):
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Milan, Lombardy
- Japan (10):
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Kuala Lumpur, Malaysia
- Philippines (2):
  - GSK Investigational Site, Makati City
  - GSK Investigational Site, Quezon City
- Poland (4):
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Mysłowice
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Łańcut
- Romania (7):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Galati
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Timișoara
- Russia (8):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kaliningrad
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Красноярск
- GSK Investigational Site, Singapore, Singapore
- South Africa (6):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Ennerdale, Gauteng
  - GSK Investigational Site, Lenasia Johannesburg, Gauteng
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Kwaguqa Emalahleni, Mpumalanga
  - GSK Investigational Site, Vosloorus Ext 2
- South Korea (6):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Ulsan
- Spain (6):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
- Taiwan (2):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Taichung
- Thailand (4):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Phitsanulok
  - GSK Investigational Site, Songkhla
- United Kingdom (3):
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Plymouth

REFERENCES:
- [Background] Yuen MF, Lim SG, Plesniak R, Tsuji K, Janssen HLA, Pojoga C, Gadano A, Popescu CP, Stepanova T, Asselah T, Diaconescu G, Yim HJ, Heo J, Janczewska E, Wong A, Idriz N, Imamura M, Rizzardini G, Takaguchi K, Andreone P, Arbune M, Hou J, Park SJ, Vata A, Cremer J, Elston R, Lukic T, Quinn G, Maynard L, Kendrick S, Plein H, Campbell F, Paff M, Theodore D; B-Clear Study Group. Efficacy and Safety of Bepirovirsen in Chronic Hepatitis B Infection. N Engl J Med. 2022 Nov 24;387(21):1957-1968. doi: 10.1056/NEJMoa2210027. Epub 2022 Nov 8. PMID 36346079
- [Derived] Joshi S, Freudenberg JM, Singh JM, Jordan WT, Felton L, Dixon S, Paff M, Theodore D, Walker J. Immunomodulation by bepirovirsen may induce killing of infected hepatocytes (B-Together study). Hepatol Int. 2025 Oct 3. doi: 10.1007/s12072-025-10917-0. Online ahead of print. PMID 41042426
- [Derived] Cremer J, Elston R, Campbell FM, Kendrick S, Paff M, Quinn G, Theodore D. B-Clear Phase 2b Study Design: Establishing the Efficacy and Safety of Bepirovirsen in Patients with Chronic Hepatitis B Virus Infection. Adv Ther. 2023 Sep;40(9):4101-4110. doi: 10.1007/s12325-023-02531-z. Epub 2023 Jul 1. PMID 37393402

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 457 participants were enrolled in the study. These 457 participants were from 2 different set of populations (referred here after as on nucleos(t)ide [NA] and not on NA therapy). Participants from these subpopulations were randomized in a ratio of 3:3:3:1 into 4 treatment arms for each population (total of 8 arms).
Groups:
- GSK3228836 for 24 Weeks (WK) (on NA Therapy): All participants of this arm received 300 milligram (mg) GSK3228836 once/week for 24 weeks (plus a loading dose of 300 mg GSK3228836 on Day 4 and 11).
- GSK3228836 for 12+12 WK (on NA Therapy); GSK3228836 for 12+12 WK (Not on NA Therapy): All participants of this arm received 300 mg GSK3228836 once/week for 12 weeks (plus a loading dose of 300 mg GSK3228836 on Day 4 and 11) followed by step-down in dose of 150 mg (plus placebo to match to maintain participant blinding) GSK3228836 once/week for 12 weeks.
- GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy); GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy): All participants of this arm received 300 mg GSK3228836 once/week for 12 weeks (plus a loading dose of 300 mg GSK3228836 on Day 4 and 11) followed by placebo once/week for 12 weeks.
- Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy); Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy): All participants of this arm received Placebo once/week for 12 weeks (plus placebo loading doses to match on Day 4 and 11) followed by 300 mg GSK3228836 once/week for 12 weeks.
- GSK3228836 for 24 WK (Not on NA Therapy): All participants of this arm received 300 mg GSK3228836 once/week for 24 weeks (plus a loading dose of 300 mg GSK3228836 on Day 4 and 11).
Period: Overall Study
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
Started | 68 | 68 | 68 | 23 | 70 | 68 | 68 | 24
Completed | 65 | 65 | 66 | 22 | 64 | 66 | 63 | 24
Not Completed | 3 | 3 | 2 | 1 | 6 | 2 | 5 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 1 | 5 | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy) | Total
Number analyzed (Participants) | 68 | 68 | 68 | 23 | 70 | 68 | 68 | 24 | 457
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 49.0 (11.54) | 46.1 (12.60) | 47.4 (11.18) | 49.8 (11.21) | 44.5 (11.10) | 43.8 (9.92) | 40.7 (11.10) | 42.4 (12.02) | 42.9 (10.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 17 | 6 | 37 | 27 | 29 | 13 | 168
  Male | 48 | 49 | 51 | 17 | 33 | 41 | 39 | 11 | 289
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 36 | 35 | 36 | 12 | 37 | 44 | 38 | 12 | 250
  Black or African American | 2 | 1 | 4 | 0 | 9 | 4 | 6 | 1 | 27
  Mixed Race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 30 | 32 | 26 | 11 | 24 | 20 | 24 | 11 | 178

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Sustained Virologic Response (SVR)
Description: The SVR was a composite endpoint defined as Hepatitis B surface antigen (HBsAg) and Hepatitis B virus (HBV) Deoxyribonucleic acid (DNA) levels were less than (<) Lower limit of quantitation (LLOQ) at the planned end of GSK3228836 treatment which is sustained for 24 weeks post-GSK3228836 treatment in the absence of rescue medication.
Time Frame: Up to Week 48
Population: The analysis was performed on the Intent to Treat (ITT) Set that includes all randomized participants who received a treatment randomization number. This population was based on the treatment the participant was randomized to. The analysis was conducted separately for the on NA treatment and not currently on NA treatment populations.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
Number analyzed (Participants) | 68 | 68 | 68 | 23 | 70 | 68 | 68 | 24
Participants | 6 | 6 | 2 | 0 | 7 | 4 | 1 | 0

2. Secondary Outcome: Number of Participants Achieving HBsAg and HBV DNA<LLOQ
Description: Participants achieving HBsAg and HBV DNA levels <LLOQ at the end of treatment (EOT) were reported.
Time Frame: Up to Week 26
Population: The analysis was performed on the ITT Set that includes all randomized participants who received a treatment randomization number. This population was based on the treatment the participant was randomized to. The analysis was conducted separately for the on NA treatment and not currently on NA treatment populations.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
Number analyzed (Participants) | 68 | 68 | 68 | 23 | 70 | 68 | 68 | 24
Participants | 16 | 9 | 8 | 4 | 17 | 10 | 6 | 1

3. Secondary Outcome: Number of Participants With Categorical Changes From Baseline in HBsAg Values
Description: Participants who achieved a decline in HBsAg values from baseline were reported. Participants were categorized in the following categorical HBsAg decline of <0.5, greater than or equal to (>=) 0.5, >=1, >=1.5, and >=3 log10 international units per milliliter (IU/mL).
Time Frame: At Baseline and Week 24
Population: The analysis was performed on the ITT set that includes all randomized participants who received a treatment randomization number. This population was based on the treatment the participant was randomized to. The analysis was conducted separately for the on NA treatment and not currently on NA treatment populations. One participant from 12+12 weeks on NA therapy arm was randomized in error and is in ITT population but did not contribute any lab data so is not part of the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
Number analyzed (Participants) | 68 | 68 | 68 | 23 | 70 | 68 | 68 | 24
Participants
  HBsAg< LLOQ, at baseline: number analyzed (Participants) | 68 | 67 | 68 | 23 | 70 | 68 | 68 | 24
  HBsAg< LLOQ, at baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HBsAg decline <0.5 log10 IU/mL: number analyzed (Participants) | 64 | 63 | 63 | 22 | 63 | 63 | 58 | 23
  HBsAg decline <0.5 log10 IU/mL | 12 | 21 | 37 | 4 | 8 | 14 | 29 | 8
  HBsAg decline >=0.5 log10 IU/mL: number analyzed (Participants) | 64 | 63 | 63 | 22 | 63 | 63 | 58 | 23
  HBsAg decline >=0.5 log10 IU/mL | 52 | 42 | 20 | 17 | 55 | 48 | 22 | 15
  HBsAg decline >=1 log10 IU/mL: number analyzed (Participants) | 64 | 63 | 63 | 22 | 63 | 63 | 58 | 23
  HBsAg decline >=1 log10 IU/mL | 48 | 38 | 14 | 17 | 51 | 36 | 18 | 15
  HBsAg decline >=1.5 log10 IU/mL: number analyzed (Participants) | 64 | 63 | 63 | 22 | 63 | 63 | 58 | 23
  HBsAg decline >=1.5 log10 IU/mL | 42 | 32 | 12 | 15 | 48 | 30 | 9 | 12
  HBsAg decline >=3 log10 IU/mL: number analyzed (Participants) | 64 | 63 | 63 | 22 | 63 | 63 | 58 | 23
  HBsAg decline >=3 log10 IU/mL | 34 | 16 | 5 | 10 | 35 | 13 | 4 | 9

4. Secondary Outcome: Number of Participants With Categorical Changes From Baseline in HBV DNA Values
Description: Participants who achieved a decline in HBV DNA values from baseline were reported. Participants were categorized in the following categorical HBV DNA decline of <1, >=1, >=2, and >=3 log IU/mL.
Time Frame: At Baseline and Week 24
Population: The analysis was performed on ITT set that includes all randomized participants who received a treatment randomization number. This population was based on the treatment participant was randomized to. One participant from 12+12 weeks on NA therapy arm who was randomized in error is in ITT population but did not contribute any lab data so is not part of the analysis. One participant from 12+12 weeks not on NA therapy has no baseline data due to insufficient sample quantity at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
Number analyzed (Participants) | 68 | 68 | 68 | 23 | 70 | 68 | 68 | 24
Participants
  HBV DNA < LLOQ, at Baseline: number analyzed (Participants) | 68 | 67 | 68 | 23 | 70 | 67 | 68 | 24
  HBV DNA < LLOQ, at Baseline | 66 | 66 | 66 | 22 | 0 | 0 | 0 | 0
  HBV DNA decline <1 log10 IU/mL: number analyzed (Participants) | 62 | 60 | 60 | 20 | 59 | 63 | 58 | 23
  HBV DNA decline <1 log10 IU/mL | 2 | 0 | 0 | 0 | 3 | 12 | 21 | 3
  HBV DNA decline >=1 log10 IU/mL: number analyzed (Participants) | 62 | 60 | 60 | 20 | 59 | 63 | 58 | 23
  HBV DNA decline >=1 log10 IU/mL | 11 | 4 | 13 | 3 | 51 | 44 | 30 | 18
  HBV DNA decline >=2 log10 IU/mL: number analyzed (Participants) | 62 | 60 | 60 | 20 | 59 | 63 | 58 | 23
  HBV DNA decline >=2 log10 IU/mL | 0 | 0 | 0 | 0 | 40 | 23 | 19 | 14
  HBV DNA decline >=3 log10 IU/mL: number analyzed (Participants) | 62 | 60 | 60 | 20 | 59 | 63 | 58 | 23
  HBV DNA decline >=3 log10 IU/mL | 0 | 0 | 0 | 0 | 27 | 19 | 11 | 9

5. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) Normalization
Description: The ALT normalization (ALT≤ upper limit of normal [ULN]) over time in absence of rescue medication in participants with baseline ALT>ULN.
  Participants who achieved ALT normalization were reported.
Time Frame: At Baseline and Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
Number analyzed (Participants) | 68 | 68 | 68 | 23 | 70 | 68 | 68 | 24
Participants
  Participants with ALT > ULN, at Baseline | 6 | 7 | 6 | 2 | 20 | 20 | 21 | 9
  Participants with ALT normalization, at Week 24: number analyzed (Participants) | 6 | 7 | 6 | 2 | 18 | 19 | 19 | 9
  Participants with ALT normalization, at Week 24 | 3 | 6 | 5 | 0 | 10 | 11 | 8 | 5

6. Secondary Outcome: Median Time to ALT Normalization
Description: Time to ALT normalization (ALT≤ULN) in the absence of rescue medication in participants with baseline ALT>ULN. Numbers of participants analyzed at Week 24 include participants with baseline ALT >ULN, and are as follows for NA therapy population: n=6 in GSK3228836 for 24 WK, n= 7 in GSK3228836 for 12 WK+12 WK, n=6 in GSK3228836 for 12 WK + Placebo for 12 WK, n=2 in Placebo for 12 WK + GSK3228836 for 12 WK, respectively. The numbers of participants analyzed are as follows for the not on NA therapy population: n=20 GSK3228836 for 24 WK, n=20 in GSK3228836 for 12 WK+12 WK, n=21 in GSK3228836 for 12 WK + Placebo for 12 WK, n=9 in Placebo for 12 WK + GSK3228836 for 12 WK arm, respectively.
Time Frame: Baseline and up to Week 48
Population: The analysis was performed on the ITT Set that includes all randomized participants who received a treatment randomization number. This population was based on the treatment the participant was randomized to. The analysis was conducted separately for the on NA treatment and not currently on NA treatment populations. Only those participants with baseline ALT>ULN were analyzed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
Number analyzed (Participants) | 6 | 7 | 6 | 2 | 20 | 20 | 21 | 9
Weeks | 16.6 [1.1 to NA] — Upper limit was Not estimable (NE) due to an insufficient number of participants with events. | 4.1 [1.0 to 11.9] | 1 [1.0 to 8.1] | 7 [1.1 to NA] — Upper limit was NE due to an insufficient number of participants. | 13.4 [2.1 to NA] — Upper limit was NE due to an insufficient number of participants with events | 15.1 [4.3 to 18.1] | 10.7 [5.1 to 21.1] | 18.1 [1 to 32.1]

7. Secondary Outcome: Number of Participants With Positive Hepatitis B Virus E-antibody (HBeAb)
Description: Blood samples were collected to assess HBeAb level and participants with positive HBeAb were reported.
Time Frame: Up to Week 48
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
Number analyzed (Participants) | 68 | 68 | 68 | 23 | 70 | 68 | 68 | 24
Participants | 3 | 4 | 5 | 2 | 6 | 4 | 6 | 3

8. Secondary Outcome: Mean HBsAg and HBV DNA Level
Description: Blood samples were collected from participants to assess HBsAg and HBV DNA level at indicated time points.
Time Frame: At Baseline, Week 12, and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Log10 (IU/mL)
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
Number analyzed (Participants) | 68 | 68 | 68 | 23 | 70 | 68 | 68 | 24
Log10 (IU/mL)
  HBsAg, at Baseline: number analyzed (Participants) | 68 | 67 | 68 | 23 | 70 | 68 | 68 | 24
  HBsAg, at Baseline | 3.29 (0.623) | 3.26 (0.608) | 3.33 (0.588) | 3.43 (0.435) | 3.72 (0.771) | 3.64 (0.721) | 3.66 (0.675) | 3.76 (0.789)
  HBsAg, at Week 12: number analyzed (Participants) | 65 | 65 | 65 | 22 | 64 | 63 | 61 | 24
  HBsAg, at Week 12 | 1.20 (1.878) | 1.04 (1.858) | 1.76 (1.706) | 3.36 (0.431) | 1.39 (1.965) | 1.27 (2.000) | 1.57 (1.808) | 3.68 (0.798)
  HBsAg, at Week 24: number analyzed (Participants) | 64 | 63 | 63 | 22 | 63 | 63 | 58 | 23
  HBsAg, at Week 24 | 0.65 (1.939) | 1.45 (1.809) | 2.51 (1.536) | 0.83 (1.801) | 0.77 (2.016) | 1.88 (1.915) | 2.88 (1.511) | 1.64 (2.171)
  HBV DNA, at Baseline: number analyzed (Participants) | 68 | 67 | 68 | 23 | 70 | 67 | 68 | 24
  HBV DNA, at Baseline | 0.48 (0.638) | 0.39 (0.603) | 0.53 (0.659) | 0.40 (0.622) | 5.02 (1.527) | 5.14 (1.557) | 4.67 (1.497) | 5.57 (1.654)
  HBV DNA, at Week 12: number analyzed (Participants) | 65 | 63 | 61 | 22 | 64 | 62 | 60 | 23
  HBV DNA, at Week 12 | 0.74 (0.654) | 0.86 (0.700) | 0.67 (0.785) | 0.61 (0.682) | 3.00 (2.242) | 2.92 (2.142) | 2.68 (1.996) | 4.96 (2.074)
  HBV DNA, at Week 24: number analyzed (Participants) | 62 | 60 | 60 | 20 | 59 | 63 | 58 | 23
  HBV DNA, at Week 24 | 0.55 (0.654) | 0.56 (0.649) | 0.56 (0.714) | 0.79 (0.667) | 2.37 (2.137) | 2.93 (2.317) | 3.07 (1.938) | 3.04 (2.224)

9. Secondary Outcome: Mean Values of Hepatitis B Virus e Antigen (HBeAg) Level
Description: Blood samples were collected from participants to assess HBeAg level at indicated time points. Participants with presence of HBeAg at baseline were analyzed at indicated timepoint. Note: The units are on the log10 scale so negative values are expected (e.g. 0.933 U/mL = -0.03 log10 U/mL).
Time Frame: At Baseline, Week 12, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log10 unit per milliliter (U/mL)
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
Number analyzed (Participants) | 18 | 20 | 24 | 7 | 21 | 16 | 16 | 7
Log10 unit per milliliter (U/mL)
  HBeAg, at Baseline | 0.49 (1.014) | 0.12 (0.756) | 0.36 (1.053) | 0.63 (1.323) | 2.13 (1.564) | 2.52 (0.919) | 1.77 (1.612) | 2.84 (0.743)
  HBeAg, at Week 12: number analyzed (Participants) | 18 | 18 | 21 | 7 | 19 | 16 | 13 | 7
  HBeAg, at Week 12 | 0.06 (1.027) | -0.21 (0.732) | 0.19 (1.089) | 0.60 (1.310) | 1.84 (1.805) | 1.52 (1.831) | 1.07 (1.551) | 2.79 (0.725)
  HBeAg, at Week 24: number analyzed (Participants) | 16 | 18 | 23 | 7 | 18 | 16 | 13 | 7
  HBeAg, at Week 24 | -0.41 (0.635) | -0.48 (0.752) | -0.19 (1.071) | 0.08 (1.497) | 1.18 (2.064) | 1.34 (1.936) | 0.89 (1.667) | 1.06 (2.165)

10. Secondary Outcome: Mean Change From Baseline in HBsAg and HBV DNA Level
Description: Blood samples were collected from participants to assess HBsAg and HBV DNA level at indicated time points. Note: The units are on the log10 scale so negative values are expected (e.g. 0.933 IU/mL = -0.03 log10 IU/mL).
Time Frame: At Baseline, Week 12, and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log IU/mL
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
Number analyzed (Participants) | 68 | 68 | 68 | 23 | 70 | 68 | 68 | 24
log IU/mL
  HBsAg, at Baseline: number analyzed (Participants) | 68 | 67 | 68 | 23 | 70 | 68 | 68 | 24
  HBsAg, at Baseline | 3.29 (0.623) | 3.26 (0.608) | 3.33 (0.588) | 3.43 (0.435) | 3.72 (0.771) | 3.64 (0.721) | 3.66 (0.675) | 3.76 (0.789)
  HBsAg, at Week 12: number analyzed (Participants) | 65 | 65 | 65 | 22 | 64 | 63 | 61 | 24
  HBsAg, at Week 12 | -2.09 (1.649) | -2.23 (1.597) | -1.59 (1.474) | -0.03 (0.089) | -2.37 (1.585) | -2.41 (1.562) | -2.06 (1.638) | -0.08 (0.292)
  HBsAg, at Week 24: number analyzed (Participants) | 64 | 63 | 63 | 22 | 63 | 63 | 58 | 23
  HBsAg, at Week 24 | -2.62 (1.653) | -1.81 (1.488) | -0.83 (1.248) | -2.57 (1.671) | -2.96 (1.656) | -1.77 (1.489) | -0.77 (1.108) | -2.09 (1.764)
  HBV DNA, at Baseline: number analyzed (Participants) | 68 | 67 | 68 | 23 | 70 | 67 | 68 | 24
  HBV DNA, at Baseline | 3.29 (0.623) | 3.26 (0.608) | 3.33 (0.588) | 3.43 (0.435) | 3.72 (0.771) | 3.64 (0.721) | 3.66 (0.675) | 3.76 (0.789)
  HBV DNA, at Week 12: number analyzed (Participants) | 65 | 63 | 61 | 22 | 64 | 61 | 60 | 23
  HBV DNA, at Week 12 | 0.24 (0.793) | 0.47 (0.773) | 0.16 (0.942) | 0.19 (0.727) | -1.96 (1.365) | -2.22 (1.592) | -1.92 (1.349) | -0.54 (1.421)
  HBV DNA, at Week 24: number analyzed (Participants) | 62 | 60 | 60 | 20 | 59 | 62 | 58 | 23
  HBV DNA, at Week 24 | 0.06 (0.831) | 0.17 (0.661) | 0.09 (0.928) | 0.33 (0.928) | -2.66 (1.646) | -2.2 (1.68) | -1.52 (1.637) | -2.6 (2.001)

11. Secondary Outcome: Mean Change From Baseline in HBeAg Level
Description: as for outcome 9
Time Frame: At Baseline, Week 12, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Log u/mL
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
Number analyzed (Participants) | 18 | 20 | 24 | 7 | 21 | 16 | 16 | 7
Log u/mL
  HBeAg, at Baseline | 0.49 (1.014) | 0.12 (0.756) | 0.36 (1.053) | 0.63 (1.323) | 2.13 (1.564) | 2.52 (0.919) | 1.77 (1.612) | 2.84 (0.743)
  HBeAg, at Week 12: number analyzed (Participants) | 18 | 19 | 24 | 7 | 18 | 16 | 13 | 7
  HBeAg, at Week 12 | -0.52 (0.874) | -0.42 (0.480) | -0.33 (0.343) | -0.17 (0.453) | -0.65 (0.919) | -1.25 (1.522) | -0.94 (1.618) | -0.14 (0.313)
  HBeAg, at WeeK 24: number analyzed (Participants) | 16 | 18 | 23 | 7 | 18 | 16 | 13 | 7
  HBeAg, at WeeK 24 | -0.85 (1.071) | -0.56 (0.811) | -0.46 (0.595) | -0.56 (0.598) | -1.01 (1.426) | -1.18 (1.532) | -0.70 (1.673) | -1.78 (2.057)

12. Secondary Outcome: Mean Hepatitis B Virus Surface Antigen Antibody (Anti-HBsAg) Level
Description: Blood samples were collected to assess anti-HBsAg level at indicated timepoints.
Time Frame: At Baseline, Week 36, and 48
Population: The analysis was performed on ITT set that includes all randomized participants who received a treatment randomization number. This population was based on the treatment participant was randomized to. One participant from 12+12 weeks on NA therapy arm who was randomized in error is in ITT population but did not contribute any lab data so is not part of the analysis. Four participants across other arms had missing anti-HBsAg baseline data.
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
Number analyzed (Participants) | 68 | 68 | 68 | 23 | 70 | 68 | 68 | 24
Log10 IU/mL
  At baseline: number analyzed (Participants) | 68 | 67 | 67 | 23 | 69 | 67 | 67 | 24
  At baseline | 0.67 (0.289) | 0.65 (0.165) | 0.64 (0.129) | 0.66 (0.287) | 0.65 (0.284) | 0.69 (0.303) | 0.62 (0.150) | 0.74 (0.307)
  At Week 36: number analyzed (Participants) | 65 | 64 | 65 | 22 | 63 | 66 | 61 | 24
  At Week 36 | 0.94 (0.534) | 0.83 (0.401) | 0.74 (0.333) | 0.79 (0.368) | 1.01 (0.660) | 0.82 (0.385) | 0.74 (0.347) | 0.90 (0.437)
  At Week 48: number analyzed (Participants) | 65 | 65 | 66 | 22 | 62 | 65 | 63 | 24
  At Week 48 | 0.88 (0.471) | 0.77 (0.368) | 0.70 (0.277) | 0.75 (0.326) | 0.91 (0.567) | 0.79 (0.369) | 0.71 (0.296) | 0.83 (0.356)

13. Secondary Outcome: Mean Change From Baseline in Anti-HBsAg Level
Description: Blood samples were collected to assess anti-HBsAg level at indicated timepoints.
Time Frame: At Baseline, Week 12, and 24
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
Number analyzed (Participants) | 68 | 68 | 68 | 23 | 70 | 68 | 68 | 24
Log10 IU/mL
  At Baseline: number analyzed (Participants) | 68 | 67 | 67 | 23 | 69 | 67 | 67 | 24
  At Baseline | 0.67 (0.289) | 0.65 (0.165) | 0.64 (0.129) | 0.66 (0.287) | 0.65 (0.284) | 0.69 (0.303) | 0.62 (0.150) | 0.74 (0.307)
  At Week 12: number analyzed (Participants) | 65 | 64 | 64 | 22 | 63 | 66 | 60 | 24
  At Week 12 | 0.28 (0.481) | 0.18 (0.343) | 0.11 (0.319) | 0.13 (0.250) | 0.37 (0.615) | 0.13 (0.353) | 0.12 (0.221) | 0.16 (0.355)
  At Week 24: number analyzed (Participants) | 65 | 65 | 65 | 22 | 62 | 65 | 62 | 24
  At Week 24 | 0.22 (0.429) | 0.12 (0.335) | 0.07 (0.267) | 0.09 (0.239) | 0.26 (0.507) | 0.10 (0.319) | 0.09 (0.203) | 0.09 (0.203)

14. Secondary Outcome: Mean Area Under the Concentration-time Curve From Time 0 up to 24 Hours (AUC0-24h) of GSK3228836
Description: Intensive pharmacokinetic (PK) sampling was done in a subset of participants on stable NA therapy to analyze AUC0-24h of GSK3228836.
Time Frame: Up to Week 24
Population: The analysis was performed on the PK Set that includes all participants in the Safety population who received an active study treatment and had at least 1 non-missing PK assessment (NQ values were considered as non-missing values).
Measure: Mean (Standard Deviation); unit: hour*micrograms per milliliter (h*ug/mL)
Groups:
- GSK3228836 Dose Level 150mg: Represents Pharmacokinetic (PK) set of participants who received GSK3228836 at a dose level of 150 mg once a week.
- GSK3228836 Dose Level 300mg: Represents Pharmacokinetic (PK) set of participants who received GSK3228836 at a dose level of 300 mg once a week.
Arm/Group | GSK3228836 Dose Level 150mg | GSK3228836 Dose Level 300mg
Number analyzed (Participants) | 12 | 12
hour*micrograms per milliliter (h*ug/mL) | 55.214 (22.9901) | 140.312 (37.3548)

15. Secondary Outcome: Mean Maximum Observed Concentration (Cmax) of GSK3228836
Description: Intensive PK sampling was done in a subset of participants on stable NA therapy to analyze Cmax of GSK3228836.
Time Frame: Up to Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- GSK3228836 Dose Level 150mg: Represents PK set of participants who received GSK3228836 at a dose level of 150 mg once a week.
- GSK3228836 Dose Level 300mg: Represents PK set of participants who received GSK3228836 at a dose level of 300 mg once a week.
Arm/Group | GSK3228836 Dose Level 150mg | GSK3228836 Dose Level 300mg
Number analyzed (Participants) | 12 | 12
ug/mL | 6.112 (2.8112) | 14.956 (5.6592)

16. Secondary Outcome: Median Time of Maximum Observed Concentration (Tmax) of GSK3228836
Description: Intensive PK sampling was done in a subset of participants on stable NA therapy to analyze tmax of GSK3228836.
Time Frame: Up to Week 24
Population: as for outcome 14
Measure: Median (Full Range); unit: hour
Arm/Group | GSK3228836 Dose Level 150mg | GSK3228836 Dose Level 300mg
Number analyzed (Participants) | 12 | 12
hour | 3.008 [2.00 to 4.02] | 3.017 [2.00 to 5.00]

17. Secondary Outcome: Mean AUC0-24h of NA Therapies
Description: Intensive PK sampling was done in a subset of participants on stable NA therapy to analyze AUC0-24h. Participants on NA therapy were stratified as per the following NA therapy Tenofovir disoproxil fumarate 245 or 300 mg once daily, Tenofovir alafenamide 25 mg once a daily or every 2 days, and Entecavir 0.5 mg once daily.
Time Frame: Up to Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: h*nanograms per milliliter (h*ng/mL)
Groups:
- Tenofovir Disoproxil Fumarate: Participants who received Tenofovir disoproxil fumarate 245 or 300 mg once daily.
- Tenofovir Alafenamide: Participants who received Tenofovir alafenamide 25 mg once daily or every 2 days.
- Entecavir: Participants who received Entecavir 0.5 mg once a daily.
Arm/Group | Tenofovir Disoproxil Fumarate | Tenofovir Alafenamide | Entecavir
Number analyzed (Participants) | 7 | 5 | 16
h*nanograms per milliliter (h*ng/mL) | 2753.908 (661.3392) | 308.167 (104.8297) | 24.43 (6.761)

18. Secondary Outcome: Mean Ctau of NA Therapies
Description: Intensive PK sampling was done in a subset of participants on stable NA therapy to analyze Ctau. Participants on NA therapy were stratified as per the following NA therapy Tenofovir disoproxil fumarate 245 or 300 mg once daily, Tenofovir alafenamide 25 mg once a daily or every 2 days, and Entecavir 0.5 mg once daily.
Time Frame: Up to Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tenofovir Disoproxil Fumarate | Tenofovir Alafenamide | Entecavir
Number analyzed (Participants) | 7 | 5 | 16
ng/mL | 57.04 (17.0787) | 10.31 (3.4802) | 0.478 (0.1055)

19. Secondary Outcome: Mean Cmax of NA Therapies
Description: Intensive PK sampling was done in a subset of participants on stable NA therapy to analyze Cmax. Participants on NA therapy were stratified as per the following NA therapy Tenofovir disoproxil fumarate 245 or 300 mg once daily, Tenofovir alafenamide 25 mg once a daily or every 2 days, and Entecavir 0.5 mg once daily.
Time Frame: Up to Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Entecavir: Participants who received Entecavir in 0.5 mg once daily.
Arm/Group | Tenofovir Disoproxil Fumarate | Tenofovir Alafenamide | Entecavir
Number analyzed (Participants) | 7 | 5 | 16
ng/mL | 318.857 (95.94) | 19.36 (5.85) | 6.526 (2.27)

20. Secondary Outcome: Median Tmax of NA Therapies
Description: Intensive PK sampling was done in a subset of participants on stable NA therapy to analyze tmax. Participants on NA therapy were stratified as per the following NA therapy Tenofovir disoproxil fumarate 245 or 300 mg once daily, Tenofovir alafenamide 25 mg once a daily or every 2 days, and Entecavir 0.5 mg once daily.
Time Frame: Up to Week 24
Population: as for outcome 14
Measure: Median (Full Range); unit: hour
Arm/Group | Tenofovir Disoproxil Fumarate | Tenofovir Alafenamide | Entecavir
Number analyzed (Participants) | 7 | 5 | 16
hour | 1 [0.52 to 1.47] | 1.417 [0.93 to 1.55] | 0.983 [0.48 to 2.02]

21. Secondary Outcome: Median Terminal Half-life (t1/2) of GSK3228836
Description: Blood samples were collected from all participants for t1/2 analysis of GSK3228836. Note: for this endpoint data for more comparable arms GSK3228836 for 24WK and 12+12 WK from both on NA and not on NA therapy were presented.
Time Frame: Up to Week 48
Population: as for outcome 14
Measure: Median (Full Range); unit: Day
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy)
Number analyzed (Participants) | 68 | 67 | 70 | 67
Day | 28.897 [7.52 to 191.98] | 24.918 [8.84 to 216.43] | 27.846 [10.19 to 149.74] | 38.205 [6.87 to 161.83]

22. Secondary Outcome: Mean Ctau of GSK3228836
Description: Blood samples were collected from all participants for Ctau analysis of GSK3228836 at indicated. Note: for this endpoint data for more comparable arms GSK3228836 for 24WK and 12+12 WK from both on NA and not on NA therapy were presented.
Time Frame: Up to Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy)
Number analyzed (Participants) | 68 | 67 | 70 | 67
ng/mL
  At Week 8: number analyzed (Participants) | 62 | 62 | 67 | 65
  At Week 8 | 21.009 (9.6214) | 47.039 (198.1345) | 21.663 (14.4479) | 23.46 (16.6498)
  At Week 12: number analyzed (Participants) | 66 | 64 | 63 | 65
  At Week 12 | 23.162 (11.8963) | 23.234 (11.6993) | 21.777 (9.9248) | 22.789 (11.7361)
  At Week 24: number analyzed (Participants) | 64 | 61 | 63 | 64
  At Week 24 | 31.102 (28.7535) | 18.95 (14.6513) | 28.158 (17.0606) | 20.138 (19.023)

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) and serious adverse events (SAEs) were collected from the signing of the informed consent until the final follow-up visit, up to 48 weeks.
Description: The safety population included participants who received at least one dose of study treatment.
  The safety population was comprised of 455 participants, 2 participants excluded from arms GSK3228836 300mg for 12 weeks in both on NA and not on NA therapy population, respectively. Both participants did not receive study treatment, one due to randomization error (on NA therapy) and other due to the participant decision due to concern of potential side effects (not on NA therapy).
Arm/Group | GSK3228836 for 24 Weeks (WK) (on NA Therapy) | GSK3228836 for 12+12 WK (on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) | GSK3228836 for 24 WK (Not on NA Therapy) | GSK3228836 for 12+12 WK (Not on NA Therapy) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy)
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/67 | 0/68 | 0/23 | 0/70 | 0/67 | 0/68 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/68 | 1/67 | 4/68 | 0/23 | 6/70 | 2/67 | 3/68 | 0/24
Other Adverse Events (participants affected / at risk) | 56/68 | 59/67 | 53/68 | 16/23 | 65/70 | 60/67 | 61/68 | 19/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3228836 for 24 Weeks (WK) (on NA Therapy) (N=68) | GSK3228836 for 12+12 WK (on NA Therapy) (N=67) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) (N=68) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) (N=23) | GSK3228836 for 24 WK (Not on NA Therapy) (N=70) | GSK3228836 for 12+12 WK (Not on NA Therapy) (N=67) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) (N=68) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy) (N=24)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cryoglobulinaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3228836 for 24 Weeks (WK) (on NA Therapy) (N=68) | GSK3228836 for 12+12 WK (on NA Therapy) (N=67) | GSK3228836 for 12 WK + Placebo for 12 WK (on NA Therapy) (N=68) | Placebo for 12 WK + GSK3228836 for 12 WK (on NA Therapy) (N=23) | GSK3228836 for 24 WK (Not on NA Therapy) (N=70) | GSK3228836 for 12+12 WK (Not on NA Therapy) (N=67) | GSK3228836 for 12 WK + Placebo for 12 WK (Not on NA Therapy) (N=68) | Placebo for 12 WK + GSK3228836 for 12 WK (Not on NA Therapy) (N=24)
Abnormal clotting factor (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 1 (1) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (6) | 2 (2) | 1 (3) | 0 (0) | 5 (9) | 2 (2) | 3 (5) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0)
Dyschromatosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Noninfective conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 4 (5) | 2 (5) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 3 (4) | 3 (3) | 3 (4) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 7 (9) | 4 (5) | 2 (2) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 5 (6) | 1 (3) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 7 (11) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 4 (6) | 1 (2) | 1 (1) | 5 (5) | 2 (2) | 3 (4) | 0 (0)
Energy increased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (8) | 4 (4) | 7 (13) | 1 (1) | 13 (19) | 7 (15) | 8 (11) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 0 (0)
Injection site anaesthesia (General disorders) | 1 (2) | 3 (8) | 2 (4) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 0 (0)
Injection site bruising (General disorders) | 7 (36) | 11 (17) | 7 (23) | 4 (13) | 13 (42) | 10 (29) | 14 (33) | 4 (10)
Injection site discolouration (General disorders) | 8 (22) | 9 (65) | 14 (92) | 2 (3) | 13 (39) | 11 (46) | 6 (37) | 2 (4)
Injection site discomfort (General disorders) | 2 (13) | 9 (62) | 9 (54) | 1 (2) | 4 (13) | 6 (25) | 4 (25) | 2 (2)
Injection site erosion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 36 (216) | 37 (175) | 34 (194) | 5 (22) | 34 (264) | 30 (150) | 37 (179) | 10 (23)
Injection site haematoma (General disorders) | 5 (9) | 3 (15) | 1 (3) | 1 (2) | 8 (17) | 4 (12) | 2 (3) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site hypoaesthesia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 3 (14) | 3 (6) | 4 (13) | 0 (0) | 6 (20) | 7 (16) | 2 (5) | 1 (1)
Injection site nodule (General disorders) | 1 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (4)
Injection site pain (General disorders) | 11 (45) | 15 (59) | 21 (118) | 6 (16) | 20 (198) | 13 (61) | 14 (66) | 6 (41)
Injection site pruritus (General disorders) | 14 (88) | 17 (78) | 15 (100) | 2 (3) | 23 (198) | 16 (85) | 19 (98) | 2 (4)
Injection site swelling (General disorders) | 4 (45) | 4 (12) | 13 (70) | 1 (2) | 10 (69) | 7 (44) | 5 (13) | 0 (0)
Injection site warmth (General disorders) | 1 (2) | 5 (13) | 2 (2) | 0 (0) | 2 (39) | 1 (34) | 4 (19) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 3 (3) | 3 (4) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 10 (14) | 6 (8) | 10 (19) | 6 (7) | 15 (23) | 17 (38) | 17 (23) | 4 (5)
Scar inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 2 (2) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Immunodeficiency (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Type III immune complex mediated reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 8 (8) | 5 (5) | 1 (1) | 3 (3) | 6 (6) | 4 (4) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes dermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 2 (2) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 0 (0) | 0 (0)
Injection site abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site cellulitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 5 (5) | 4 (4) | 4 (6) | 2 (2) | 4 (6) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pustule (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 3 (4) | 2 (2) | 1 (1)
Urethritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 4 (4) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (3) | 0 (0)
Vaginitis gardnerella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 2 (2) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post vaccination syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth avulsion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 2 (2) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (13) | 8 (10) | 4 (6) | 5 (5) | 17 (25) | 15 (18) | 12 (21) | 4 (9)
Albumin urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Antineutrophil cytoplasmic antibody positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Antinuclear antibody positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 8 (11) | 9 (12) | 7 (9) | 2 (4)
Autoantibody positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubin conjugated increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Complement factor C3 decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 7 (8) | 4 (5) | 6 (6) | 4 (4)
Complement factor C4 decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 4 (5) | 4 (4) | 3 (3)
Complement factor abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complement factor increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 1 (1) | 4 (4) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 2 (4) | 6 (21) | 1 (2) | 1 (1) | 1 (1) | 2 (10) | 1 (3) | 2 (3)
Creatinine urine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Crystal urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hepatitis B DNA assay positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immature granulocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mean cell volume decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 4 (6) | 0 (0) | 2 (2) | 1 (1) | 8 (11) | 3 (6) | 3 (3) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Total complement activity decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary sediment present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urine albumin/creatinine ratio (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (15) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (4) | 6 (8) | 1 (1) | 1 (1) | 3 (6) | 4 (5) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (5) | 6 (8) | 0 (0) | 4 (6) | 4 (4) | 3 (5) | 2 (2)
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (6) | 4 (4) | 0 (0) | 10 (12) | 7 (10) | 2 (2) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (4) | 0 (0) | 4 (4) | 3 (6) | 2 (2) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 3 (3) | 4 (6) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (10) | 6 (8) | 8 (15) | 3 (3) | 14 (25) | 14 (50) | 14 (26) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Albuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cylindruria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 2 (3) | 1 (2)
Ketonuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Nephrocalcinosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (3) | 2 (3) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 3 (3) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 2 (3) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asteatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 2 (2) | 2 (6) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (6) | 2 (2) | 1 (2) | 1 (1) | 5 (5) | 4 (12) | 3 (7) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (8) | 1 (7) | 1 (1) | 0 (0) | 1 (1) | 7 (11) | 5 (13) | 1 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (4) | 2 (2) | 0 (0)
Urticarial vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular pain (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT04449029/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/29/NCT04449029/SAP_001.pdf